CLINICAL TRIAL: NCT04414761
Title: A Randomized Control Trial to Compare the Live Birth Rate Between the Progestin-primed Ovarian Stimulation Protocol and the GnRH Antagonist Protocol in Patients With Anticipated High Ovarian Response Undergoing IVF
Brief Title: Live Birth Rate Between PPOS and GnRH Antagonist Protocol in Patients With Anticipated High Ovarian Response
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JIAI 2020-06
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-03

CONDITIONS: IVF; GnRH Antagonist; PPOS
MeSH Terms: interventions — Progesterone; Medroxyprogesterone; Dydrogesterone; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; cetrorelix; ganirelix

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antagonist group (Active Comparator): Women will receive antagonist (Cetrorelix or Ganirelix 0.25mg) once subcutaneously daily from day 6 of ovarian stimulation till the day of the ovulation trigger.
  Interventions: Drug: GnRH Antagonist
- PPOS group (Experimental): Women will receive oral medroxyprogesterone 10 mg daily or duphaston 10mg bd daily from Day 3 till the day of ovulation trigger.
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — oral medroxyprogesterone 10 mg daily or duphaston 10mg bd daily from Day 3 till the day of ovulation trigger
  Other Names: medroxyprogesterone; duphaston
  Arms: PPOS group
Drug: GnRH Antagonist — GnRH antagonist (Cetrorelix or Ganirelix 0.25mg) once subcutaneously daily from day 6 of ovarian stimulation till the day of the ovulation trigger
  Other Names: Cetrorelix; Ganirelix
  Arms: Antagonist group

SUMMARY:
Progestin can inhibit the pituitary LH surge during ovarian stimulation and various studies show progestin-primed ovarian stimulation (PPOS) is effective in blocking the LH surge in IVF. More and more centers in China are using PPOS because this regimen appears simpler and cheaper.A randomized trial to compare the effectiveness of PPOS and GnRH antagonist protocol in IVF in terms of the live birth rate is urgently needed.

Trial objectives: To compare the live birth rate between the PPOS protocol and the antagonist protocol used for ovarian stimulation during IVF

Eligible women will be randomised into one of the two groups:

Antagonist group : Women will receive antagonist (Cetrorelix or Ganirelix 0.25mg) once subcutaneously daily from day 6 of ovarian stimulation till the day of the ovulation trigger.

PPOS group: Women will receive oral medroxyprogesterone 10 mg daily or duphaston 10mg bd daily from Day 3 till the day of ovulation trigger.

There will be no fresh transfer. Only one blastocyst will be allowed to replaced in the first FET and a maximum of two blastocysts will be replaced in the subsequent FET cycles.

The primary outcome is the live birth rate of the first frozen-thawed transfer cycle.

ELIGIBILITY:
Inclusion Criteria:

* Age of women <43 years at the time of ovarian stimulation for IVF
* The first IVF cycle
* Antral follicle count (AFC) >15 on day 2-5 of the period

Exclusion Criteria:

* Presence of a functional ovarian cyst with E2>100 pg/mL
* Recipient of oocyte donation
* Undergoing preimplantation genetic testing
* Presence of hydrosalpinx or endometrial polyp which is not surgically treated

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 784 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
live birth rate | deliveries ≥22 weeks gestation with heartbeat and breath
  live birth rate of the first frozen embryo transfer cycle

SECONDARY OUTCOMES:
positive serum hCG | 2 weeks after FET
  serum β-hCG ≥10 mIU/mL of the first FET
clinical pregnancy | 6 weeks' gestation
  presence of intrauterine gestational sac by trans-vaginal ultrasound at 6 gestational weeks of the first FET
biochemical pregnancy | 6 weeks' gestation
  positive serum hCG not followed by clinical pregnancy of the first FET
implantation rate | 6 weeks' gestation
  the number of gestational sacs per blastocyst transferred of the first FET
ongoing pregnancy | 12 weeks' gestation
  a viable pregnancy beyond 12 weeks' gestation of the first FET
cumulative live birth | 2 years' after FET
  cumulative live birth within 6 months of randomization
number of oocytes retrieved | 1 day after oocyte retrieval
  number of oocytes retrieved
number and grading of blastocysts | 1 week after oocyte retrieval
  number and grading of blastocysts suitable for biopsy and freezing
multiple pregnancy | multiple pregnancy beyond gestation 12 weeks
  more than one intrauterine sacs on scanning
ectopic pregnancy | ectopic pregnancy during 12 weeks gestation
  pregnancy outside the uterine cavity
birthweight of newborns | 1 year after FET
  the birth weight of newborns
serum baseline FSH | day 2-3 of period
  baseline FSH of period day 2-3
estradiol level on the trigger day | 2 days before oocyte retrieval
progesterone level on the trigger day | 2 days before oocyte retrieval
estradiol and progesterone levels in the follicular fluid | 1 year after FET
  estradiol and progesterone levels in the follicular fluid
miscarriage | 22 weeks of pregnancy
  clinically recognised pregnancy loss before 22 weeks of pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: XIAOXI SUN, PHD, Study Director — Shanghai JiAi Genetics & IVF Institute
Locations (1):
- ShangHai JIAI Genetics&IVF Institute, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results after deidentification (text, tables, figures, and appendices) and study protocol will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available when beginning 3 months and ending 5 years following article publication.
Access Criteria: To achieve aims in the approved proposal, researchers who provide a methodologically sound proposal will be shared with. Proposals should be sent to lihe198900@163.com.

REFERENCES:
- [Background] Begueria R, Garcia D, Vassena R, Rodriguez A. Medroxyprogesterone acetate versus ganirelix in oocyte donation: a randomized controlled trial. Hum Reprod. 2019 May 1;34(5):872-880. doi: 10.1093/humrep/dez034. PMID 30927417
- [Background] Yu S, Long H, Chang HY, Liu Y, Gao H, Zhu J, Quan X, Lyu Q, Kuang Y, Ai A. New application of dydrogesterone as a part of a progestin-primed ovarian stimulation protocol for IVF: a randomized controlled trial including 516 first IVF/ICSI cycles. Hum Reprod. 2018 Feb 1;33(2):229-237. doi: 10.1093/humrep/dex367. PMID 29300975
- [Background] Massin N. New stimulation regimens: endogenous and exogenous progesterone use to block the LH surge during ovarian stimulation for IVF. Hum Reprod Update. 2017 Mar 1;23(2):211-220. doi: 10.1093/humupd/dmw047. PMID 28062551
- [Background] Kuang Y, Chen Q, Fu Y, Wang Y, Hong Q, Lyu Q, Ai A, Shoham Z. Medroxyprogesterone acetate is an effective oral alternative for preventing premature luteinizing hormone surges in women undergoing controlled ovarian hyperstimulation for in vitro fertilization. Fertil Steril. 2015 Jul;104(1):62-70.e3. doi: 10.1016/j.fertnstert.2015.03.022. Epub 2015 May 5. PMID 25956370
- [Background] Dong J, Wang Y, Chai WR, Hong QQ, Wang NL, Sun LH, Long H, Wang L, Tian H, Lyu QF, Lu XF, Chen QJ, Kuang YP. The pregnancy outcome of progestin-primed ovarian stimulation using 4 versus 10 mg of medroxyprogesterone acetate per day in infertile women undergoing in vitro fertilisation: a randomised controlled trial. BJOG. 2017 Jun;124(7):1048-1055. doi: 10.1111/1471-0528.14622. PMID 28276192
- [Background] Alexandru P, Cekic SG, Yildiz S, Turkgeldi E, Ata B. Progestins versus GnRH analogues for pituitary suppression during ovarian stimulation for assisted reproductive technology: a systematic review and meta-analysis. Reprod Biomed Online. 2020 Jun;40(6):894-903. doi: 10.1016/j.rbmo.2020.01.027. Epub 2020 Feb 5. PMID 32327297
- [Derived] Chen ZQ, Ai A, Zhang Y, Li H, Wang JY, Wang L, Ng EHY. A randomized controlled trial to compare the live birth rate of the first frozen embryo transfer following the progestin-primed ovarian stimulation protocol vs. the antagonist protocol in women with an anticipated high ovarian response. Fertil Steril. 2024 Jun;121(6):937-945. doi: 10.1016/j.fertnstert.2024.01.027. Epub 2024 Jan 23. PMID 38272383